CLINICAL TRIAL: NCT03725735
Title: Group Cognitive Behavioral Therapy for Problem Gambling with a Focus on Emotion Regulation - a Pilot Study
Brief Title: Emotion Regulation Group Treatment for Gambling Disorder - a Pilot Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Anne H Berman, associate Professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017/1479-31/1
Record Dates: First submitted 2018-08-21; First posted 2018-10-31 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Gambling Disorder
Keywords: Gambling disorder; psychiatric comorbidities; emotion regulation
MeSH Terms: conditions — Gambling; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: Open label pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CBT for PG with emotion regulation (Experimental): A new treatment protocol for problem gamblers, CBT for problem gambling with emotion regulation, has a focus on emotion regulation, a component that has been lacking in current published research.
  Interventions: Behavioral: CBT for problem gambling with emotion regulation

INTERVENTIONS:
Behavioral: CBT for problem gambling with emotion regulation — CBT group treatment for problem gambling with emotion regulation focus, with 8 sessions.

SUMMARY:
Group cognitive behavioral therapy for Gambling Disorder (GD) with a focus on emotion regulation - A pilot study This pilot study will evaluate the feasibility and possible effectiveness of a novel treatment protocol developed within the research group including emotion regulation techniques for the treatment of GD.

DETAILED DESCRIPTION:
The manual is based on principles from so called third wave cognitive behavioral therapy, which differs from current treatment within standard care in that focus is more on emotion regulation techniques. The treatment consists of an 8- session program delivered by weekly sessions. The study is an open trial in order to evaluate the possible benefit of components of emotion regulation in treating gambling disorder (GD). Participants with psychiatric comorbidities will be included and symptoms of comorbidities will be measured as secondary outcomes.

Once included in the study the participant will be measured weekly on symptoms of gambling disorder.

By increasing competencies in emotion regulation (such as active problem solving, acceptance and reappraisal of events in order to change their emotional impact) the hypothesis is that the participants will improve on measures of symptoms of GD as well as gambling expenditure in terms of time and money.

ELIGIBILITY:
Inclusion Criteria:

* Gambling Disorder according to DSM 5

Exclusion Criteria:

* Unable to speak and read Swedish
* Symptoms of manic episode
* Severe psychiatric condition in need of urgent care

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in gambling symptoms | Pre-treatment up to 12-month followup.
  Change in gambling symptoms will be measured by Gambling symptoms assessment scale (G-SAS) - a 12-item scale measuring symtoms of gambling disorder within the last week. Maximum score 48. Higher scores indicating more severe problems.
Change in gambling expenditure | Pre-treatment up to 12-month followup.
  Change in time and money spent on gambling, per week

SECONDARY OUTCOMES:
Symptoms of depression | PHQ-9 will be administered: assessment prior to treatment, weekly measures during the 8 weeks of treatment, at treatment termination and 3, 6 and 12 months after treatment termination.
  Patient health questionnaire, PHQ-9 - measuring symtoms of depression with the last 2 weeks. Maximum score: 27. Higher scores indicating more severe problems.
Symptoms of anxiety | GAD- 7 will be administered: assessment prior to treatment, weekly measures during the 8 weeks of treatment, at treatment termination and 3, 6 and 12 months after treatment termination.
  Generalized Anxiety Disorder 7 item, GAD-7.Maximum score: 21. Higher scores indicating more severe problems
WHOQOL-Bref | WHOQOL-Bref will be administered: assessment prior to treatment, at treatment termination and 3, 6 and 12 months after treatment termination.
  Measures quality of life in four domains (psychological, social, environmental and physical)

OTHER OUTCOMES:
Gambling Urges | will be administered: assessment prior to treatment, at treatment termination and 3, 6 and 12 months after treatment termination.
  Gambling Urge Scale, 6 item - measuring gambling urges. Maximun score of 18. Higher score = stronger urges.
Craving experiences | CEQ-G will be administered: assessment prior to treatment, at treatment termination and 3, 6 and 12 months after treatment termination.
  Craving experiences questionnaire for gambling (CEQ-G)- measuring gambling cravings in terms of frequency and intensity within the last week. 16 item scores from 0-10. Maximum score of 160. Higher scores = more strong and/or intense cravings.
Alcohol consumption | AUDIT will be administered: assessment prior to treatment, at treatment termination and 3, 6 and 12 months after treatment termination.
  Alcohol Use Disorder Identification Test, AUDIT
Drug consumption | DUDIT will be administered: assessment prior to treatment, at treatment termination and 3, 6 and 12 months after treatment termination.
  Drug Use Disorder Identification Test, DUDIT
Increased competencies in Emotion Regulation | DERS - 16 will be administered: assessment prior to treatment, at treatment termination and 3, 6 and 12 months after treatment termination.
  Difficulties in Emotion Regulation Scale, DERS- 16
Increased psychological flexibility | AAQ-II will be administered: assessment prior to treatment, weekly measures during the 8 weeks of treatment, at treatment termination and 3, 6 and 12 months after treatment termination.
  Acceptance and Action Questionnaire - AAQ - II - a measure of psychological flexibility and acceptance which will be analysed as mediator in treatment. 6 items, maximum score of 42. Higher scores indicating more inflexibility and experiential avoidance.

CONTACTS AND LOCATIONS:
Overall Officials: Anne H Berman, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Center for Psychiatry Research, Karolinska Institutet, Stockholm, Sweden

REFERENCES:
- [Background] Mansson V, Molander O, Carlbring P, Rosendahl I, Berman AH. Emotion regulation-enhanced group treatment for gambling disorder: a non-randomized pilot trial. BMC Psychiatry. 2022 Jan 6;22(1):16. doi: 10.1186/s12888-021-03630-3. PMID 34991511